CLINICAL TRIAL: NCT00973375
Title: Angiographic and Intravascular Ultrasound (IVUS) Follow-up After Simultaneously Implanted Different Drug-eluting Stents in Same Individuals
Acronym: AIFSIDDES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liuhuaqiao Hospital (Other)
Responsible Party: Dingcheng Xiang, MD., Ph.D, Liuhuaqiao Hospital
Other Study IDs: LHQ09-003
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Drug Eluting Stent
Keywords: Drug-eluting stent; coronary restenosis; coronary thrombosis
MeSH Terms: conditions — Coronary Restenosis; Coronary Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endeavor group and Excel group: Endeavor group: measurements from the vessels implanted Endeavor stent(s). Excel group: measurements from the vessels implanted Excel stent(s).

SUMMARY:
The purpose of this study is to investigate if there is any different follow-up results by angiography and IVUS between two different drug-eluting stents after implanted simultaneously in same individuals.

ELIGIBILITY:
Inclusion Criteria:

* These patients who received two kinds of drug-eluting stent (Endeavor and Excel) im simultaneously.

Exclusion Criteria:

* Dual anti-platelet therapy less than 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These patients who received two kinds of drug-eluting stent (Endeavor and Excel) im simultaneously.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-05

PRIMARY OUTCOMES:
Segment and instent restenosis measured by coronary angiography and IVUS. | at 12 months after implantation

SECONDARY OUTCOMES:
Uncovered and malposition of stent. | at 12 months after implantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Liuhuaqiao Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Waseda K, Miyazawa A, Ako J, Hasegawa T, Tsujino I, Sakurai R, Yock PG, Honda Y, Kandzari DE, Leon MB, Fitzgerald PJ; ENDEAVOR IV Trial Investigators. Intravascular ultrasound results from the ENDEAVOR IV trial: randomized comparison between zotarolimus- and paclitaxel-eluting stents in patients with coronary artery disease. JACC Cardiovasc Interv. 2009 Aug;2(8):779-84. doi: 10.1016/j.jcin.2009.05.015. PMID 19695548
- [Background] Lee CH, Zhang J, Kailasam A, Tai BC, Ye F, Low AF, Hou X, Hay ET, Teo SG, Lim YT, Chen S, Tan HC. An intravascular ultrasound study of Cypher, Taxus, and endeavor stents on relation between neointimal proliferation and residual plaque burden. J Interv Cardiol. 2008 Dec;21(6):519-27. doi: 10.1111/j.1540-8183.2008.00397.x. Epub 2008 Oct 21. PMID 18973509
- [Background] Miyazawa A, Ako J, Hongo Y, Hur SH, Tsujino I, Courtney BK, Hassan AH, Kandzari DE, Honda Y, Fitzgerald PJ; ENDEAVOR III Investigators. Comparison of vascular response to zotarolimus-eluting stent versus sirolimus-eluting stent: intravascular ultrasound results from ENDEAVOR III. Am Heart J. 2008 Jan;155(1):108-13. doi: 10.1016/j.ahj.2007.08.008. Epub 2007 Sep 14. PMID 18082499